CLINICAL TRIAL: NCT01652326
Title: Clinical Quality Improvement of Benzodiazepine-Resistant Alcohol Withdrawal Syndrome
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: UPittsburgh 0031860
Record Dates: First submitted 2012-07-20; First posted 2012-07-30 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Alcohol Withdrawal Syndrome
MeSH Terms: interventions — Diazepam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Benzodiazepine-resistant: those patients with either 1) a requirement of either 200 mg of diazepam (or diazepam equivalents) in 4 hrs; 2) >40mg of diazepam (or diazepam equivalents) in 1 hr; or 3) an individual dose of 40 mg or greater of intravenous diazepam for control of agitation
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Diazepam

SUMMARY:
The overarching goal of this project is to improve the clinical quality of patients with Benzodiazepine-resistant alcohol withdrawal syndrome.

ELIGIBILITY:
Inclusion Criteria:

either

1. a requirement of either 200 mg of diazepam (or diazepam equivalents) in 4 hrs;
2. > 40mg of diazepam (or diazepam equivalents) in 1 hr; or
3. an individual dose of 40 mg or greater of intravenous diazepam for control of agitation

Exclusion Criteria:

* if < 18 years of age or had evidence of use of other illicit substances as determined by urine toxicology screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized inpatients
Sampling Method: Non-Probability Sample
Enrollment: 792 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Identify those risk factors predictive of benzodiazepine-resistant alcohol withdrawal syndrome | up to 38 months

SECONDARY OUTCOMES:
Drug utilization of phenobarbital, propofol, dexmedetomidine, and ketamine in benzodiazepine-resistant alcohol withdrawal syndrome | Up to 38 months
  Will compare the frequency, duration and dosages of the above agents when used for benzodiazepine-resistant alcohol withdrawal
Effectiveness of phenobarbital, propofol, dexmedetomidine, and ketamine in benzodiazepine-resistant alcohol withdrawal | Up to 38 months
  Comparative markers will include:
  1. Presence or absence of the following: delirium tremens, hallucinosis, seizures, or arrhythmias
  2. Indication and duration of mechanical intubation
  3. Nosocomial infection rates
  4. ICU length of stay
Tolerability of phenobarbital, propofol, dexmedetomidine, and ketamine in benzodiazepine-resistant alcohol withdrawal | Up to 38 months
  Comparative markers will include:
  1. Rikers Sedation Scale Assessments
  2. Hypotension
  3. Hypertriglyceridemia/Pancreatitis
  4. Drug induced hallucinosis or seizures

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States